CLINICAL TRIAL: NCT05764343
Title: Investigation of the Effectiveness of Immediate Smoking Cessation Interventions During Routine Outpatient Service in Current Smoker Chronic Airway Disease Patients
Brief Title: The Effect of Immediate Smoking Cessation Interventions for Smokers With Chronic Airway Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Turkish Thoracic Society (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Associated Professor Doctor, MD, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKGG
Record Dates: First submitted 2023-02-11; First posted 2023-03-10 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Tobacco Cessation; Asthma COPD; Bronchiectasis Adult
Keywords: tobacco cessation; asthma; COPD; bronchiectasis; immediate cessation support
MeSH Terms: conditions — Tobacco Use Cessation; Asthma; Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine support/care arm (No Intervention): As the followed routine implementation, this group will be given a brief smoking cessation intervention and will be recommended to apply to smoking cessation outpatient clinics by getting an appointment from quit services.
- Immediate support arm (Active Comparator): Those randomized to this group will have an immediate appointment at the smoking cessation outpatient clinic in addition to the brief smoking cessation intervention.
  Interventions: Other: Immediate smoking cessation support

INTERVENTIONS:
Other: Immediate smoking cessation support — Smoker patients with chronic airway diseases (asthma and/or COPD and/or bronchiectasis) will be evaluated for the inclusion criteria. Afterwards they will be randomized as routine support arm (as the current procedure of the care) and immediate support arm (intensive brief cessation advices following by the immediate arrangement of the appointment from the same clinic's smoking cessation service). Both arms will be followed remotely at first week and third months of the randomization regarding their quit status as well as their use of evidence based cessation treatments.
  Arms: Immediate support arm

SUMMARY:
Smoking cessation support is provided by smoking cessation outpatient clinics in our country. Smokers with chronic airway diseases can also apply to these services by making an appointment from quit lines. Quit rates of that group patients were found to be similar to the general population. In novel smoking cessation support approaches immediate cessation support is reported to be more effective than routine practice. The sample in these studies consists of individuals who applied for lung health screening programmes. There is no study in the literature examining the effect of this immediate support on patients with chronic airway diseases' quit success. Our aim with this study is to examine impact of immediate cessation support by getting an appointment to the same cessation clinic instantly on our sample's cessation success.

DETAILED DESCRIPTION:
Patients who are current smokers (who have smoked at least 100 cigarettes in their lifetime and still smoke daily or some days) will be randomized in a 1:1 ratio to the two arms in sequential order of presentation, after they have been identified and given written informed consent about the study. Demographic and clinical features will be filled. A brief smoking cessation intervention will be applied to one group and they will be recommended to apply to smoking cessation outpatient clinics by obtaining appointment from quit lines, as the way of current routine practice. Those randomized to the other group will have an immediate appointment at the smoking cessation outpatient clinic in addition to the brief smoking cessation intervention. Both patient groups will be called after 1 week by phone to inquire about their smoking cessation status and their application to smoking cessation outpatient clinics. Both groups will be called again in the 3rd month and their smoking cessation status, their application to smoking cessation outpatient clinics, and the duration/status of using pharmacological smoking cessation treatments will be questioned.

ELIGIBILITY:
Inclusion Criteria:

1. Being age 18 years and over,
2. Having diagnoses of asthma and/or COPD and/or bronchiectasis for at least 6 months,
3. Applying to the chest diseases outpatient clinics,
4. Being an current smoker,
5. Those who agree to participate in the study,
6. Patients who can be reached by phone calls at 1 week and 3 months after randomization.

Exclusion Criteria:

1. Those with active psychiatric disorders
2. Patients with impaired cognitive functions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Quit rate of both study arms | At third month of randomization
  To compare the quit rate at third month of randomization in the both arms: intensive support arm compared to routine support arm. A quitter will be considered who have never smoked since the target quit day.

SECONDARY OUTCOMES:
Smoking cessation outpatient clinic application rate of both study arms | At third month
  The admission status to smoking cessation outpatient clinics of both arms will be evaluated: admitted at least once or never admitted.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Karadoğan, Principal Investigator — Recep Tayyip Erdogan University
Locations (1):
- Recep Tayyip Erdoğan University, Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jimenez-Ruiz CA, Andreas S, Lewis KE, Tonnesen P, van Schayck CP, Hajek P, Tonstad S, Dautzenberg B, Fletcher M, Masefield S, Powell P, Hering T, Nardini S, Tonia T, Gratziou C. Statement on smoking cessation in COPD and other pulmonary diseases and in smokers with comorbidities who find it difficult to quit. Eur Respir J. 2015 Jul;46(1):61-79. doi: 10.1183/09031936.00092614. Epub 2015 Apr 16. PMID 25882805
- [Result] Karadogan D, Onal O, Kanbay Y. How does reimbursement status affect smoking cessation interventions? A real-life experience from the Eastern Black Sea region of Turkey. Tob Induc Dis. 2019 Jan 22;17:05. doi: 10.18332/tid/100412. eCollection 2019. PMID 31582917
- [Result] Williams PJ, Philip KEJ, Gill NK, Flannery D, Buttery S, Bartlett EC, Devaraj A, Kemp SV, Addis J, Derbyshire J, Chen M, Morris K, Laverty AA, Hopkinson NS. Immediate, Remote Smoking Cessation Intervention in Participants Undergoing a Targeted Lung Health Check: Quit Smoking Lung Health Intervention Trial, a Randomized Controlled Trial. Chest. 2023 Feb;163(2):455-463. doi: 10.1016/j.chest.2022.06.048. Epub 2022 Aug 4. PMID 35932889
- [Result] Buttery SC, Williams P, Mweseli R, Philip KEJ, Sadaka A, Bartlett EJ, Devaraj A, Kemp S, Addis J, Derbyshire J, Chen M, Morris K, Laverty A, Hopkinson NS. Immediate smoking cessation support versus usual care in smokers attending a targeted lung health check: the QuLIT trial. BMJ Open Respir Res. 2022 Feb;9(1):e001030. doi: 10.1136/bmjresp-2021-001030. PMID 35121633
- [Derived] Karadogan D, Telatar TG, Kaya I, Atli S, Kabil NK, Marim F, Senel MY, Yuksel A, Yalcin B, Gultekin O, Ercelik M, Akgun M. Immediately scheduled for an appointment to smoking cessation clinics: Key to quitting smoking in chronic airway disease - a multicenter randomized study. Tob Induc Dis. 2025 Jun 5;23. doi: 10.18332/tid/204254. eCollection 2025. PMID 40475312